CLINICAL TRIAL: NCT00446433
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled,Parallel-Group Study to Evaluate the Safety and Efficacy of CC-5013 in the Treatment of Adolescents and Adults With Moderately Severe Crohn's Disease
Brief Title: A Study to Evaluate CC-5013 in the Treatment of Adolescents and Adults With Moderately Severe Crohn's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CC-5013-CD-001
Record Dates: First submitted 2007-03-07; First posted 2007-03-12 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Lenalidomide

INTERVENTIONS:
Drug: CC-5013

SUMMARY:
A Multicenter, Randomized, Double-Blind, Placebo-Controlled,Parallel-Group Study to Evaluate the Safety and Efficacy of CC-5013 in the Treatment of Adolescents and Adults with Moderately Severe Crohn's Disease

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects > 12 and < 75 years of age.
2. Adolescent and adult female subjects must be of non-childbearing potential (hysterectomy) or be using one highly effective method (e.g., IUD, hormonal contraception, tubal ligation) of birth control during the entire study. Abstinence will be considered an acceptable method of birth control for adolescent females aged 12-17 years who are not sexually active and who the investigator feels will be compliant with this requirement for the 12-week treatment period. Female subjects who are post-menopausal must have had 24 continuous months of amenorrhea.
3. Negative pregnancy test for females of child bearing potential.
4. A history of Crohn's Disease (CD) of greater than 1-year duration diagnosed and documented by standard clinical, radiographic, endoscopic, histopathological criteria.
5. Signs and symptoms of moderately severe CD as defined by a Crohn's Disease Activity Index (CDAI) score of > 220 and < 400.
6. Normal thyroid function as documented by normal TSH (thyroid stimulating hormone).
7. The subject's treatment for CD must be unchanged, as described below:

   The start date of the medications listed below must be at least 4 weeks prior to randomization, and the dose must have been unchanged for at least 2 weeks prior to that visit. Medication doses may be decreased but not increased throughout the study. If not currently using these agents, the stop date of any previous treatment with these agents must be at least 4 weeks prior to randomization. The medications are:
   * oral or systemic corticosteroids
   * metronidazole (Flagyl®)
   * sulfasalazine
   * oral mesalamine
   * oral olsalazine
   * topical rectal therapy with corticosteroids or mesalamine
8. The start date of the medications listed below must be at least 3 months (12 weeks) prior to randomization, and the dose must have been unchanged for at least 4 weeks. Medication doses may be decreased but not increased throughout the study. If not currently using these agents, the stop date of any previous treatment with these agents must be at least 6 weeks prior to randomization. The medications are:

   * azathioprine (AZA)
   * 6-mercaptopurine (6 MP)
   * methotrexate
9. Subject's screening laboratory test results must meet the following criteria:

   * hemoglobin > 8.5 g/dL.
   * white blood cells (WBC) > 3.5 x 109 / L.
   * neutrophils > 1.5 x 109/L and lymphocytes >0.5 x 109/L.
   * platelets > 100 x 109 / L.
   * bilirubin, alanine transaminase (ALT), aspartate transaminase (AST) , and alkaline phosphate levels must not be above two times the upper limit of the normal range.
   * serum albumin > 3.2 mg /dL for adults (18-75) and serum albumin > 2.8 mg/dL for adolescents between the ages of 12-17.
   * serum creatinine < 2.0 mg/dL
10. Subjects must be able to adhere to the study visit schedule and other protocol requirements.
11. The subject must understand and voluntarily sign an informed consent document. Adolescent subjects under 18 years of age must have parent/guardian consent as evidenced by a signature on the consent form as well as their own assent, as evidenced by signature on the consent form.
12. The subject must be at least 25 kg (55 lbs).

Exclusion Criteria:

1. Pregnancy or lactation.
2. Predisposition to cardiac arrhythmias and history of clinically significant cardiac disease.
3. Diagnosis of ulcerative colitis.
4. CD that is limited to the stomach and proximal small intestine.
5. Known severe fixed symptomatic stenosis or stricture of the small or large intestine.
6. Current evidence of bowel obstruction, or history within the 3 months preceding randomization confirmed with objective radiographic or endoscopic evidence of a stricture with resulting obstruction (dilation of the bowel proximal to the stricture observed upon barium enema or an inability to traverse the stricture at endoscopy.
7. Subjects who have undergone a proctocolectomy or total colectomy with ileorectal anastomosis; segmental colectomy is permitted.
8. Colostomy or ileostomy.
9. Subjects with fulminant disease requiring parenteral steroid treatment, hospitalization, or felt to be in imminent need of surgery, i.e. toxic megacolon, active gastrointestinal bleeding, history of significant ulcer disease and/or esophagitis, peritonitis, intestinal obstruction, perforation, or intra-abdominal abscess requiring surgical drainage.
10. Subjects requiring intravenous nutritional support with total parenteral nutrition (TPN)/partial parenteral nutrition (PPN) that provides > 50 % of total daily caloric intake.
11. Subjects in whom enteral nutrition with elemental or semi-elemental formula comprises more than 50% of their total daily caloric intake. For adolescents between the ages of 12-17, subjects in whom enternal nutrition with elemental or semi-elemental formula comprises more the 75% of their total daily caloric intake.
12. Current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, hematological, endocrine (including thyroid as documented by an abnormal TSH), pulmonary, cardiac, neurological, or cerebral disease, including the following specific exclusions: uncontrolled diabetes, unstable ischemic heart disease, uncontrolled or recent seizures, autoimmune diseases not related to inflammatory bowel diseases, chronic respiratory insufficiency, or recent cerebral vascular accident (within 2 months of randomization).
13. Serious infections or history of opportunistic infections; less serious infections within 3 months of randomization, such as acute upper respiratory tract infections (colds) or uncomplicated urinary tract infection are permitted at the discretion of the Investigator. The following are specific exclusions:

    * Chronic hepatitis B and C
    * Documented HIV infection, ARC (AIDS related complex), AIDS, or immune deficiency.
14. Stool examination positive for enteric pathogens (including Clostridium difficile),pathogenic ova, or parasites.
15. Concomitant or recent medication use as follows:

    * Treatment with any other therapeutic agent targeted at reducing TNF-a, e.g., CC-1088, thalidomide, cyclosporine, or pentoxifylline within 4 weeks of randomization, and mycophenolate (Cellcept), infliximab (Remicadeä), Enbrelä, or FK506 (Tacrolimus) within 8 weeks of randomization
    * Treatment with interleukin-2 or -10 or other immunomodifier agent within 24 weeks of randomization.
    * Requirement of systemic corticosteroid therapy for other disease(s), e.g., asthma. Inhaled steroids for treating asthma are acceptable for this protocol.
    * Subjects receiving anticoagulant therapy (other than a total daily aspirin dose of 325 mg or less).
    * Subjects having received non CD-directed antibiotic therapy within 2 weeks of randomization. CD-directed antibiotic therapy, for example with ciprofloxacin or metronidazole, is acceptable provided the dose has been stable for the 2 weeks prior to randomization.
    * Subjects who have received an investigational drug within 30 days of randomization.
16. Subjects with a history of malignancy, except basal cell or squamous cell carcinoma of the skin or cervical carcinoma in situ.
17. Dysplasia (low-grade or high-grade) of the colon/small bowel within the last 5 years prior to screening.
18. Subjects who, in the judgment of the Investigator, are unwilling or unable to comply with all the protocol-related assessments and procedures, including completion of a daily diary.
19. History of alcohol or other drug abuse within 1 year of randomization, or any conditions associated with poor compliance.
20. Subjects in whom multiple venipunctures are not feasible due to poor tolerability or lack of easy access.
21. Any condition which, in the opinion of the Investigator, places the subject at unacceptable risk if he/she were to participate in the study.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90
Dates: Start 2002-03; Study Completion 2003-12

CONTACTS AND LOCATIONS:
Locations (18):
- United States (5):
  - Advanced Clinical Therapeutics, Tucson, Arizona
  - Advanced Clinical Research Institute, Anaheim, California
  - Washington Hospital Center Physicians Office Building, Washington D.C., District of Columbia
  - Springfield Clinic, Springfield, Illinois
  - Wake Research Associates, Raleigh, North Carolina
- Hopital Saint Louis, Paris, France
- Israel (3):
  - Rambam Hospital, Haifa
  - Department of Medicine A, Liver & Gastroenterology Units, Jerusalem
  - Department of Gastroenterology and Hepatology, Tel Litwinsky
- United Kingdom (9):
  - Department of Gastroenterology, Dartford, Kent
  - Department of Gastroenterology, Bristol
  - Addenbrookes Hospital, Cambridge
  - Department of Medicine, Cardiff
  - Department of Gastroenterology, London
  - Department of Gastroenterology, Manchester
  - St. Mark's Hospital, Middlesex
  - Department of Gastroentroerology, Newcastle
  - Nottingham

REFERENCES:
- [Background] Mansfield JC, Parkes M, Hawthorne AB, Forbes A, Probert CS, Perowne RC, Cooper A, Zeldis JB, Manning DC, Hawkey CJ. A randomized, double-blind, placebo-controlled trial of lenalidomide in the treatment of moderately severe active Crohn's disease. Aliment Pharmacol Ther. 2007 Aug 1;26(3):421-30. doi: 10.1111/j.1365-2036.2007.03385.x. PMID 17635377